CLINICAL TRIAL: NCT05801900
Title: Intravenous Ibuprofen Versus Ketorolac for Perioperative Pain Control in Morbid Obese Patients Undergoing Bariatric Surgery: a Randomized Controlled Trial
Brief Title: Intravenous Ibuprofen Versus Ketorolac in Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-340-2022
Record Dates: First submitted 2023-03-13; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain; Bariatric Surgery Candidate
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketorolac group (Active Comparator): ketorolac 30 mg (diluted in 200 mL normal saline) intravenously over 5 minutes
  Interventions: Drug: Ketorolac group
- Ibuprofen group (Active Comparator): ibuprofen 800 mg intravenously (Diluted in 200 mL of normal saline) over 5 minutes
  Interventions: Drug: Ibuprofen group

INTERVENTIONS:
Drug: Ketorolac group — 30 min preoperatively then every 8 hours postoperatively
  Arms: Ketorolac group
Drug: Ibuprofen group — 30 min preoperatively then every 8 hours postoperatively
  Arms: Ibuprofen group

SUMMARY:
The aim of the current study is to compare the analgesic effects of both drugs in patients with obesity undergoing bariatric surgery.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and prophylactic antiemetic will be provided in the form of slow intravenous injection of 5 mg dexamethasone drugs.

Anesthesia Anesthesia will be induced with 2 mg/kg propofol, 2 mcg/kg fentanyl (lean body weight), and tracheal intubation will be facilitated by 0.6 mg/kg ideal body weight rocuronium after loss of consciousness. Anesthesia will be maintained with isoflurane 1-1.2% in oxygen and 0.1 mg/kg rocuronium every 30 minutes. Fentanyl boluses of 1 mcg/kg will be given if heart rate or/and systolic blood pressure >120% of baseline.

Postoperatively, pain assessments using the visual analogue scale (VAS) will be performed at rest and during movement (knee flexion) at 0.5, 4, 10, 18, and 24 h after leaving the operating room. If the VAS score is > 3 intravenous nalbuphine 0.1-0.2 mg/kg (lean body weight) titrated to response with maximum single dose of 20 mg and maximum daily dose of 160 mg.

Intravenous ondansetron 4 mg will be given to treat postoperative nausea or vomiting

ELIGIBILITY:
Inclusion Criteria:

* adult (18-65 years) patients
* body mass index ≥35 kg/m2
* scheduled for laparoscopic bariatric surgery

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical class IV,
* severe cardiac comorbidity (impaired contractility with ejection fraction < 50%, heart block, significant arrhythmias, tight valvular lesions),
* known obstructive sleep apnea or patients with STOP-bang score ≥5,
* baseline SpO2 <95%,
* renal impairment,
* allergy to any of study's drugs,
* history of gastrointestinal bleeding or ulceration, or inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
VAS | 30 minutes after extubation
  Visual analogue scale

SECONDARY OUTCOMES:
total intraoperative fentanyl | 30 seconds after skin incision until 1 min after skin closure
  mcg
post operative nalbuphine | 30 minutes after extubation until 24 hours postoperatively
  mg
VAS | at 0.5, 4, 10, 18, and 24 hours after extubation
  Visual analogue scale
time to independent movement | 30 minutes after extubation until 24 hours postoperatively
  defined as time from extubation to be able independently mobile e.g. using the bathroom

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data from this study are available from the PI upon resealable request